CLINICAL TRIAL: NCT06451042
Title: FET-PET/MRI Based Treatment Planning for Glioblastoma Multiforme in Post-Surgical Patients (FET-TREAT)
Acronym: FET-TREAT
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 5919
Record Dates: First submitted 2024-05-31; First posted 2024-06-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma Multiforme
Keywords: FET-PET; Glioblastoma; GBM; 0-(2-18F-Fluoroethyl)-L-Tyrosine (FET); Glioma
MeSH Terms: conditions — Glioblastoma; Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-Operative GBM Positron Emission Tomography/Magnetic Resonance Imaging (PET/MRI): 0-(2-18F-Fluoroethyl)-L-Tyrosine (FET) PET/MRI for planning of radiation therapy of post-operative glioblastoma multiforme patients
  Interventions: Diagnostic Test: FET-PET/MRI

INTERVENTIONS:
Diagnostic Test: FET-PET/MRI — Radiation planning target volume (PTV) when planned with FET-PET/MRI to PTV when planned with conventional (Standard of Care) MRI only. 0-(2-18F-Fluoroethyl)-L-Tyrosine (FET) 180-200 megabecquerel (MBq) administered intravenously prior to PET/MRI imaging.

SUMMARY:
Glioblastoma multiforme (GBM) represent the most common primary brain malignancy and prognosis remains poor. The most common subtype is glioblastoma which has a 5-year survival rate of approximately 5%. Despite advances in MRI techniques, accurately determining total extent of tumor remains a challenge. The result is incomplete treatment resulting in reduced survival or overtreatment resulting in avoidable treatment related morbidity. A more accurate means of assessing tumor extent is needed to guide management to improve patient survival and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Each participant must meet all of the following inclusion criteria to participate in this study:

* ≥ 18 years of age
* Diagnosis of glioblastoma multiforme
* Post-maximally safe surgical resection
* No prior radiation or systemic treatment for high grade glioma
* Able to tolerate PET/MRI scan with intravenous contrast
* Willing to provide informed consent

Exclusion Criteria:

All participants meeting any of the following exclusion criteria at baseline screening will be excluded from participation in this study:

* MRI contraindication
* Creatinine clearance < 30mL/min
* Inability to lie still for 60 minutes
* Gadolinium allergy
* Positive pregnancy test
* Breastfeeding
* Patient unable to follow the protocol for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of both males and females over 18 years of age post maximally safe resection of glioblastoma multiforme and intent to treat with stereotactic radiation.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Difference in radiation treatment volume as determined by FET-PET/MRI compared to standard of care MRI. | 12 months
  Volume difference measured in cubic centimetres

OTHER OUTCOMES:
Difference in pre- and post-treatment metabolic tumor volume as determined by FET-PET. | 12 months
  Volume difference measured in cubic centimetres
Overall and recurrence-free survival post radiation treatment. | 12 months
  Measured in months
Quality of life changes pre and post radiation treatment. | 12 months
  Units on a scale - Linear Analog Self-Assessment, score minimum = 0, score maximum = 10, higher is better

CONTACTS AND LOCATIONS:
Overall Officials: Amit Singnurkar, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT06451042/ICF_000.pdf